CLINICAL TRIAL: NCT04257123
Title: SATISFY (geleSis100 Effects on AppeTIte Sensations, Feeding Behavior and Dietary energY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Gelesis, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor of Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 055-051
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: Following an initial 3-day run-in period (feeding only), participants will be randomly assigned to two 1-week controlled feeding periods with and without Gelesis100. After a one week washout, participants will complete the other pattern. Following another 1-week washout, participants will be randomly assigned again to two 1-week free-feeding periods with and without Gelesis100. After a one week washout, participants will complete the other pattern.
Who Masked: Participant, Investigator
Masking Description: Treatment with Gelesis100 or placebo will be double-blinded and randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Controlled-Feeding (Experimental): For two weeks (separated by a wash-out week), participants will consume all meals in the Nutrition Science facility.
  Interventions: Device: Gelesis100; Other: Placebo
- Free-Feeding (Experimental): For two weeks (separated by a wash-out week), participants will receive no dietary guidance and will be allowed to consume whatever they desire.
  Interventions: Device: Gelesis100; Other: Placebo

INTERVENTIONS:
Device: Gelesis100 — Participants will administer Gelesis100 before lunch and dinner meals.
Other: Placebo — Participants will administer a placebo before lunch and dinner meals.

SUMMARY:
A recent clinical trial demonstrated the efficacy of Gelesis100 use for weight loss (Obes 2019;27:205-216). The present trial is designed to explore the mechanisms by which it may work, i.e. by suppressing hunger, altering food intake and/or altering the efficiency of energy extraction from food.

DETAILED DESCRIPTION:
Overweight/obesity is prevalent and associated with multiple adverse health outcomes. Moderating energy intake is one approach to lose or maintain body weight. To improve the probability of long-term adherence to an energy restricted diet, it is important to address the issue of appetite control. Numerous food components and properties have been explored for their satiation/satiety value. Two physical properties known to impact appetite are viscosity and elasticity (properties common to many dietary fibers). These properties may work by multiple mechanisms including prolonged gastric distention after a meal and slowed gastric emptying resulting in moderated swings in blood glucose and insulin concentrations. These properties may also alter the efficiency of energy absorption.

The present trial will test the effects of Gelesis100, a FDA cleared superabsorbent hydrogel, on the mechanisms just noted. Gelesis100 is nonsystemic and works directly in the gastrointestinal tract. Gelesis100 is made from two natural ingredients, cellulose and citric acid, that form a three-dimensional matrix designed to occupy volume in the stomach and small intestine, to create a sensation of fullness. The capsules disintegrate in the stomach and release the Gelesis100 particles, which can hydrate up to 100 times their original weight. When fully hydrated, the Gelesis100 particles occupy about a quarter of average stomach volume (although this may vary based on body size and various other factors). Without increasing the caloric value of a meal, Gelesis100 particles mix with ingested foods and create thousands of small, nonclustering individual gel pieces. The gel particles mix with ingested foods, creating a larger volume with higher elasticity and viscosity in the stomach and small intestine, promoting satiety and fullness. Gelesis100 has been cleared by FDA through the 510k de novo process and is marketed as a prescription medical device for weight management under the trade name Plenity™. A recent clinical trial demonstrated the efficacy of its use for weight loss (Obes 2019;27:205-216). The present trial is designed to explore the mechanisms by which it may work, i.e. by suppressing hunger, altering food intake and/or altering the efficiency of energy extraction from food.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years (this is to reduce the number of people who apply that are taking medications or have chronic diseases).
* BMI =25-40 kg/m2

Exclusion Criteria:

* Body weight fluctuation of >5kg in the past 3 months
* Participant is allergic to or objects to consuming CMC, Citric acid, Sodium stearyl fumarate, titanium oxide, or gelatin.
* Participants with esophageal anatomic anomalies including webs, diverticuli, and rings
* Participants with suspected strictures (such as patients with Crohn's disease)
* Participants with complications from prior gastrointestinal surgery that could affect GI transit and motility
* Participants with active gastrointestinal conditions such as gastro-esophageal reflux disease (GERD), ulcers, or heartburn
* Participants taking prescribed medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Appetite Ratings | up to 2 weeks
  Hunger, fullness, desire to eat and thirst will be measured on visual analogue scales with end anchors of "not at all" to "extremely." Ratings will be captured via Qualtrics software. Also, subjects will be asked to indicate when, during the meals, they feel full on the first and last days of the Controlled-Feeding periods.
Eating Behavior | up to 2 weeks
  A battery of validated questionnaires related to Ingestive behavior will be completed. These include Power of Food Scale, Emotional Eating Scale, Three-Factor Eating Questionnaire-Revised, Food Craving Inventory-II, Barratt Impulsiveness Scale, Adult Eating Behavior Scale, Self-Regulation of Eating Behavior Questionnaire for Adults, Meal Pattern Questionnaire, Study-Specific Appetite and Eating Behavior Questionnaire.
Dietary Assessment | up to 2 weeks
  Diet composition during the free-feeding periods will be assessed by diet histories taken by a registered dietitian through the Nutrition Assessment Center.
Fecal energy and macronutrient compostion | With initiation of each Controlled-Feeding period, participants will swallow a capsule containing a red dye. They will monitor bowel movements until the red dye is passed. All stool will be collected from this point forward.
  A quantitative stool collection method will be used. Collections will be homogenized and aliquots will be freeze-dried. Energy and macronutrient composition analysis of feces will be conducted in triplicate.

SECONDARY OUTCOMES:
Weight | up to 8 weeks
  Body weight will be measured
Compliance | up to 2 weeks
  Eighty milligrams of PABA will be taken in capsule form with the pre-lunch and pre-dinner beverage to serve as a compliance biomarker during the Free-Feeding periods. 24-hour urine samples will be collected in 3 L opaque collection bottles. Urinary PABA recovery will be analyzed using spectrophometric methods. Completeness of PABA collection will calculated as the measure of compliance ( ). Compliance will also be assessed by counting capsules returned by the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States